CLINICAL TRIAL: NCT01008761
Title: A Double Blind Randomized Control Trail of Azithromycin for the Acute Management of Wheezy Pre-school Children
Brief Title: Trial for the Treatment of Acute Asthma in Wheezy Pre-school Aged Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Janielee Williamson (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Sponsor-Investigator, Janielee Williamson, CCCRP Research Coordinator, Alberta Children's Hospital
Organization: Alberta Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALAWhZy2010
Record Dates: First submitted 2009-11-04; First posted 2009-11-06 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Asthma
Keywords: Pre-school child; Wheezy episode
MeSH Terms: conditions — Asthma | interventions — Azithromycin; Macrolides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zithromax, 100 mgmgs; 5mls suspension (Active Comparator): Azithromycin given at 10 mg/kg/day for day 1, then 5 mg/kg for 4 days Each syringe will contain 12.5 mls (250 mgs) sufficient drug to adequately dose children who with up to 25 kgs (95%tile for weight for 60 month old child)
  Interventions: Drug: Azithromycin
- Suspension placebo, (Placebo Comparator): placebo (suspension produced by CDC Edmonton.) given at 10 mg/kg/day for day 1, then 5 mg/kg for 4 days.
  Interventions: Drug: Suspension Placebo

INTERVENTIONS:
Drug: Azithromycin — Azithromycin given at 10 mg/kg/day for day 1, then 5 mg/kg for 4 days Each syringe will contain 12.5 mls (250 mgs) sufficient drug to adequately dose children who with up to 25 kgs (95%tile for weight for 60 month old child)
  Other Names: Azithromycin, zithromax, macrolide
  Arms: Zithromax, 100 mgmgs; 5mls suspension
Drug: Suspension Placebo — Placebo suspension will be administered on day 1 at 10mg/kg and then for the next 4 days at 5 mg/kg
  Other Names: Azithromycin
  Arms: Suspension placebo,

SUMMARY:
To determine if treatment of pre-school children with a history of wheeze who present to an Emergency Department with an acute wheezing episode with azithromycin for 5 days will resolve their symptoms more quickly, will require less short acting beta agonist (SABA), and allow these children to remain symptom free for a longer period of time.

ELIGIBILITY:
Inclusion Criteria:

* 12-60 months
* wheeze on auscultation

Exclusion Criteria:

* antibiotic use in the past 30 days
* macrolide allergy
* underlying medical condition
* significant co-morbidities
* current enrollment
* language barrier or no access to phone for follow up

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 440 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To determine if treatment of pre-school children with a history of wheeze who present to an Emergency department (ED) with an acute wheezing episode with Azithromycin for 5 days will resolve their symptoms more quickly | Patient is followed by phone day 1,3,5,7,14, with an in person return visit on day 21 and then by phone again every 2 weeks for 6 months

SECONDARY OUTCOMES:
Treatment of pre-school children with acute wheezing symptoms with 5 days of azithromycin will cause these children to use less rescue beta2 agonists than those treated with placebo | Patient is followed by phone day 1,3,5,7,14, with an in person return visit on day 21 and then by phone again every 2 weeks for 6 months
Treatment of pre-school children with acute wheezing symptoms with 5 days of azithromycin will allow these children to remain free of subsequent wheezy episodes longer than those treated with placebo. | Patient is followed by phone day 1,3,5,7,14, with an in person return visit on day 21 and then by phone again every 2 weeks for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David W Johnson, MD, Principal Investigator — Alberta children's Hospital/University of Calgary; Piush Mandhane, MD, Principal Investigator — Stollery Children's Hospital Edmonton
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta